CLINICAL TRIAL: NCT00323427
Title: Clinical Trial of the "Living Well With Hearing Loss Workshop"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4185-R
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-01

CONDITIONS: Hearing Loss; Stress
Keywords: Audiology; Coping behaviors; Counseling; Hearing aids; Hearing impairment; Patient-centered care; Psychological adaptation; Psychological adjustment; Rehabilitation; Social adjustment; Aural Rehabilitation
MeSH Terms: conditions — Hearing Loss; Social Adjustment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Group Aural Rehabilitation session, two hours in length, approximately 6 participants plus Group Facilitator
  Interventions: Behavioral: The Living Well with Hearing Loss Workshop; Device: hearing aid services
- Arm 2 (Active Comparator): Veterans receive new VA issued digital hearing aids per Standard VA Audiology Hearing Aid services
  Interventions: Device: hearing aid services

INTERVENTIONS:
Behavioral: The Living Well with Hearing Loss Workshop — Interactive group session modeled on Patient-Centered medicine and Adult Learning principles; the participants are partners with the Group Facilitator who is a hearing rehabilitation professional
  Arms: Arm 1
Device: hearing aid services — Standard VA audiological hearing aid dispensing services

SUMMARY:
This study evaluates whether a 2 hour group session, "The Living Well with Hearing Loss Workshop," can successfully teach hard of hearing people how to best use hearing aids and a variety of personal skills to compensate for the limitations of their impaired ears.

DETAILED DESCRIPTION:
Hearing aids are essential to the rehabilitation of veterans who have acquired hearing loss. However, as with most prosthetic devices, the use of hearing aids does not result in fully normal functioning, and research shows that residual handicapping effects of hearing loss recur for many veterans. Hearing loss now affects 31 million Americans and is increasing in prevalence due to the "graying of America" and the noise-traumas of modern life, including modern warfare. VA spent over $119,000,000 on hearing aid technology for eligible veterans in FY 2004.Therefore, evidence-based rehabilitation treatments to alleviate avoidable hearing handicaps is a priority for VA and non-VA audiology. VA audiology clinics, however, are forced by high work loads to follow tight schedules for fitting hearing aids, with little time available to counsel veterans on skills for dealing effectively with the auditory and psychosocial challenges specific to their personal life style.

The proposed study will present and evaluate a single session, two hour long rehabilitation treatment model, "The Living Well with Hearing Loss Workshop." This cost-effective group intervention draws from research in psychology and behavioral medicine, as well as audiology, to teach specific skills that empower veterans to self-manage the adverse consequences of their hearing loss. The workshops will use multi-media presentations to train participating veterans in cognitive, behavioral and affective coping skills, while the patient-centered process focuses on collaborative problem-solving of hearing-loss-challenges participants present to their groups as personally important.

This is a dual site, randomized clinical trial, conducted by Co-PIs Dr. Turbin, a psychologist and Investigator at the NCRAR in the Portland, Oregon VAMC; and Dr. Abrams, a rehabilitative audiologist and Chief of Audiology Services at the Bay Pines, Florida VAMC. We will recruit a total of 310 veterans, all patients at the VAMC audiology clinics in Portland or Bay Pines, who are: 1) recipients of their first hearing aids, 2) have a mild to moderately-severe hearing loss in their better ear, and 3) present no other condition that would preclude their participation in age-appropriate interpersonal activities. Half of these veterans will be randomized to each of our two treatments: the Control condition of routine VA hearing-aid-rehabilitation-alone, and our Experimental Treatment condition of routine audiology services plus our workshop intervention. All subjects will complete three questionnaires as Pre-test measures before hearing aid fitting, eight weeks after hearing aid fitting as Re-tests and then four months later as Post-tests. An additional personality inventory will be administered only at baseline, yielding co-variates for interpreting possible within-group variance. Workshop participants will attend their session within one month of hearing aid fitting. The workshops will be facilitated by audiologists we will train in our empowering, patient-centered, coping-skills based model.

We hypothesize that our Workshop participants will show enhanced personal adjustment and use of communication strategies when compared to both baseline and to Control subjects, and further hypothesize that our Workshop participants will exceed our Controls in self reported hearing aid benefit at Re-test, and retain these differential treatment benefits at Post-test. The outcome data will enhance our understanding about the coping processes by which people respond to their hearing disability and its treatment by hearing-aids-alone, and about how well Workshop participants learn and utilize the skills taught in our treatment model. The findings from this research can foster continued development and implementation of evidence-based rehabilitation treatments and, if shown to be effective, our model can be replicated at audiology clinics, adapted for video or online training, or used by other health care professionals or even lay mentors to enhance the quality of life of people who are hard of hearing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are users of new hearing aids with mild to severe hearing loss in better ear.

Exclusion Criteria:

* Patient has been in aural rehabilitation in the past 2 years, or has a condition besides hearing loss that affects age-appropriate social activity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel B Turbin, Principal Investigator — VA Medical Center, Portland
Locations (2):
- United States (2):
  - VA Medical Center, Bay Pines, Bay Pines, Florida
  - VA Medical Center, Portland, Portland, Oregon

REFERENCES:
- See also: Study site URL — http://www.ncrar.research.va.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Aural Rehabilitation: Group Aural Rehabilitation session, two hours in length, approximately 6 participants plus Group Facilitator
- Hearing Aids: Veterans receive new VA issued digital hearing aids per Standard VA Audiology Hearing Aid services
Period: Overall Study
Arm/Group | Group Aural Rehabilitation | Hearing Aids
Started | 69 | 66
Completed | 38 | 43
Not Completed | 31 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 69 | 66 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 20 | 53
  >=65 years | 36 | 46 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (9.8) | 71.1 (8.4) | 69.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 69 | 65 | 134
Region of Enrollment [Number; unit: participants]
  United States | 69 | 66 | 135

OUTCOME MEASURES:

1. Primary Outcome: Communication Profile for Hearing Impaired: Maladaptive Strategies Subscale
Description: The Communication Profile for Hearing Impaired (CPHI) queries subjects on how well they can communicate with others.
  The Maladaptive strategies subscale describe behaviors that prevent the individual from coping effectively with communication problems.
  8 week change score from baseline value. Larger values of the change score indicate less use of maladaptive behaviors. Larger group mean change score indicates BETTER performance on this scale.
  CPHI Maladaptive strategies subscale ranges from 1 (better) to 5 (worse) maladaptive strategy usage.
Time Frame: 8 weeks post-baseline relative to baseline
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 57 | 58
score on a scale | 0.33 (0.53) | 0.37 (0.51)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; H0: Mean(Arm 1) = Mean(Arm 2); Test type: Superiority or Other; p = 0.69, t-test, 2 sided — No multiple testing adjustment; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [-0.15 to 0.23], Standard Error of Mean 0.0974

2. Primary Outcome: Communication Profile for Hearing Impaired: Verbal Strategies Subscale
Description: The Communication Profile for Hearing Impaired (CPHI) queries subjects on how well they can communicate with others.
  The Verbal Strategies subscale describe adaptive strategies for coping with the effects of hearing impairment on communication.
  8 week change score from baseline value.
  Larger values of the change score indicate more use of adaptive Verbal Strategies.
  Larger group mean change score indicates BETTER performance on this scale.
  CPHI Verbal Strategies scores vary from 1 (worse) to 5 (best) strategy usage.
Time Frame: 8 weeks post-baseline relative to baseline
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 57 | 58
score on a scale | -0.34 (0.79) | -0.23 (0.67)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; H0: Mean(Arm 1) = Mean(Arm 2); Test type: Superiority or Other; p = 0.42, t-test, 2 sided — No adjustment; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.16 to 0.38], Standard Error of Mean 0.14

3. Primary Outcome: Communication Profile for Hearing Impaired : Non-verbal Strategies Subscale
Description: The Communication Profile for Hearing Impaired (CPHI) queries subjects on how well they can communicate with others.
  The Non-verbal Strategies subscale describe adaptive coping strategies but they describe unobtrusive, nonverbal behaviors that the individual can use to maximize communication effectiveness.
  8 week change score from baseline value.
  Larger values of the change score indicate more use of adaptive non-verbal behaviors.
  Larger group mean change score indicates BETTER performance on this scale.
  The CPHI Non-verbal strategies score ranges from 1 (worse) to 5 (better) usage of non-verbal strategies.
Time Frame: 8-weeks post-baseline relative to baseline
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: score on a scale.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 57 | 58
score on a scale. | -0.22 (0.78) | -0.22 (0.83)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; H0: mean(Arm 1) = Mean (Arm 2); Test type: Superiority or Other; p = 0.97, t-test, 2 sided — No adjustment; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.30 to 0.29], Standard Error of Mean 0.15

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/66
Other Adverse Events (participants affected / at risk) | 0/69 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes